CLINICAL TRIAL: NCT00626574
Title: A Double Blinded, Placebo Controlled, Pilot Study to Evaluate the Safety of Treating Patients With Aneurysmal SubArachnoid Hemorrhage (SAH) With Epoetin Alfa
Brief Title: Treating Patients With Aneurysmal SubArachnoid Hemorrhage (SAH) With Epoetin Alfa
Acronym: EPO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study is terminated as a result of data from a study that showed increased mortality in stroke patients.
Sponsor: University of South Florida (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: Principal Investigator, Enrico Camporesi, Emeritus Professor, Dept of Surgery, University of South Florida
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 105838c; USF 6176-P67638
Record Dates: First submitted 2008-02-07; First posted 2008-02-29 (Estimated); Results first posted 2012-10-29 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Epoetin alfa; aneurysm; subarachnoid hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm | interventions — Epoetin Alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Group A will receive Procrit® intravenous injections (40,000U) once daily for 3 days (Study Days 1, 2, and 3). The first dose of Procrit® will be given within 36 hours of the initial SAH event / symptoms and immediately before the vascular clipping procedure.
  Interventions: Drug: Epoetin alfa
- B (Placebo Comparator): Group B will receive Saline intravenous injections once daily for 3 days (Study Days 1, 2, and 3).
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Epoetin alfa — Intravenous administration of epoetin alfa (40,000 IU) immediately before clipping surgery. Successive doses will be given 24 and 48 hours after the first dose.
  Other Names: Procrit
  Arms: A
Drug: Saline — 3ml of saline will be administered via an IV push immediately before clipping surgery. Successive doses will be given 24 and 48 hours after the first dose.
  Arms: B

SUMMARY:
This is a prospective, randomized, double-blinded, placebo controlled pilot safety study that will enroll a total of twenty subjects. Subjects will be adults (30-75) who have sustained a SAH secondary to cerebral aneurysm rupture and who present with minimal neurological symptoms. All subjects will have a Hemoglobin less than or equal to 12 g/dL within 24 hours prior to study entry and undergo operative aneurismal clipping. Subjects will be randomized into two groups, ten subjects receiving the drug and ten subjects receiving the placebo. The subjects will receive three intravenous injections of study drug or placebo, once before undergoing operative aneurysmal clipping (study Day 1) and again for two additional days (study Day 2 and study Day 3).

There are 3 phases to this trial:

Screening Phase - patients will present with Subarachnoid hemorrhage (SAH) and prepped for surgery within 36 hours Treatment Phase - first pre-operative dose before surgery (Study Day 1), post-operative (Study Days 2 and 3) Follow-up Phase- Study Day 4 through discharge, 6-7 week follow-up Primary Objective: To determine the safety of administering intravenous doses of Procrit® once daily for three consecutive days to patients with aneurysmal SAH before and after vascular clipping by comparing the incidence of thrombotic events, hemoglobin and 6-7 week mortality between the Procrit® and placebo groups. Secondary Objectives: To determine if administration of Procrit® prior to aneurysm clipping reduces the incidence of vasospasm following a SAH event treated by vascular clipping. To determine if Procrit® administration prior to aneurysm clipping in patients with Aneurysmal SAH will improve neurological assessment scores in the post-SAH/post-clipping time period. To determine the feasibility of organizing a larger, randomized study to explore the neuroprotective effect of Procrit® in patients with Aneurysmal SubArachnoid Hemorrhage (SAH) when Procrit® is administered prior to surgical clipping of the aneurysm.

It is hypothesized that Procrit will provide a significant level of neuroprotection in the brain after an SAH event as a result of reduced cell death, as well as a reduced amount of vasospasm activity and delayed cerebral ischemia which can occur as a result of SAH. These factors may contribute to improved neurological functioning scores when compared to the placebo treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 30-75
* Patients undergoing vascular clipping post SAH
* Aneurysmal SAH as determined by history or clinical evaluation
* WFNS Score I and II
* Hb ≤ 12 g/dL within 36 hours prior to first dose of study drug
* Patients who receive Study drug and undergo surgical clipping of the aneurysm within 36 hours of the SAH event

Exclusion Criteria:

* Non-aneurysmal SAH
* WFNS Score III and higher
* Patients presenting with previous history of SAH
* Terminal, brain-dead, comfort care patients
* Patients not undergoing vascular clipping
* Hb > 12 g/dL
* Patients receiving blood transfusion prior to surgery
* Patients who currently receive Procrit or an EPO product
* Patients undergoing surgical clipping of the aneurysm greater than 36 hours after the SAH event
* Pregnancy or lactating
* Renal insufficiency (must present and maintain normal creatinine levels)
* Uncontrolled hypertension (systolic > 150 mmHg)
* Active or known seizure history within one year of SAH event
* Known history of thrombotic vascular events (PE, DVT, AMI, stroke)
* Allergy or sensitivity to mammalian derived products

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrico M Camporesi, MD, Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Procrit: Group A will receive Procrit® intravenous injections (40,000U) once daily for 3 days (Study Days 1, 2, and 3). The first dose of Procrit® will be given within 36 hours of the initial SAH event / symptoms and immediately before the vascular clipping procedure.
- Saline: Group B will receive Saline intravenous injections once daily for 3 days (Study Days 1, 2, and 3).
Period: Overall Study
Arm/Group | Procrit | Saline
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Procrit | Saline | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events After Administering Intravenous Doses of Procrit® Once Daily for Three Consecutive Days to Patients With Aneurysmal SAH Before and After Vascular Clipping
Description: Number of adverse events
Time Frame: First 10 days following clipping and 6 week F/U
Population: Pilot Study- per protocol
Measure: Number; unit: adverse events
Arm/Group | Procrit | Saline
Number analyzed (Participants) | 2 | 1
adverse events | 1 | 2

2. Secondary Outcome: To Determine if Administration of Procrit® Prior to Aneurysm Clipping Reduces the Incidence of Vasospasm Following a SAH Event Treated by Vascular Clipping.
Time Frame: first 10 days following clipping and 6 week f/u
Population: Study terminated prematurely. Outcome measures were not analyzed.
Groups:
- Group A: Group A will receive Procrit® intravenous injections (40,000U) once daily for 3 days (Study Days 1, 2, and 3). The first dose of Procrit® will be given within 36 hours of the initial SAH event / symptoms and immediately before the vascular clipping procedure.
  Epoetin alfa: Intravenous administration of epoetin alfa (40,000 IU) immediately before clipping surgery. Successive doses will be given 24 and 48 hours after the first dose.
- Group B: Group B will receive Saline intravenous injections once daily for 3 days (Study Days 1, 2, and 3).
  Saline: 3ml of saline will be administered via an IV push immediately before clipping surgery. Successive doses will be given 24 and 48 hours after the first dose.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: To Determine if Procrit® Administration Prior to Aneurysm Clipping in Patients With Aneurysmal SAH Will Improve Neurological Assessment Scores in the Post-SAH/Post-clipping Time Period
Time Frame: First 10 days following clipping and 6 week f/u
Population: Study was terminated prematurely and outcome measures were not analyzed.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: To Determine the Feasibility of Organizing a Larger, Randomized Study to Explore the Neuroprotective Effect of Procrit® in Patients With Aneurysmal SubArachnoid Hemorrhage (SAH) When Procrit® is Administered Prior to Surgical Clipping of the Aneurysm.
Time Frame: When all data is collected and analyzed
Population: Study was terminated prematurely and outcome measures were not analyzed.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Procrit | Saline
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/1
Other Adverse Events (participants affected / at risk) | 1/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Procrit (N=2) | Saline (N=1)
Severe Headache (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Procrit (N=2) | Saline (N=1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Pseudo aneurysm left groin (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
In late October 2008, we received a letter from the sponsor requesting that we terminate any further work on this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No